CLINICAL TRIAL: NCT06173037
Title: A Multicenter, Single-arm, Phase 2 Study to Evaluate the Efficacy, Safety and Pharmacokinetics of RC88 Monotherapy in Platinum-resistant Recurrent Epithelial Ovarian, Fallopian Tube and Primary Peritoneal Cancer
Brief Title: RC88 in Platinum-Resistant Recurrent Epithelial Ovarian Cancer, Fallopian Tube Cancer, and Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC88-C008
Record Dates: First submitted 2023-11-29; First posted 2023-12-15 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Primary Peritoneal Cancer; Fallopian Tube Cancer; Epithelial Ovarian Cancer
Keywords: Primary Peritoneal Cancer; Fallopian Tube Cancer; Epithelial Ovarian Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC88 for Injection (Experimental): Participants will receive RC88 2.0 mg/kg every 3 weeks (Q3W)
  Interventions: Drug: RC88

INTERVENTIONS:
Drug: RC88 — 2.0 mg/kg Q3W IV
  Other Names: RC88 for Injection

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and pharmacokinetics of RC88 monotherapy in subjects with Platinum-Resistant Recurrent Epithelial Ovarian, Fallopian Tube and Primary Peritoneal Cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to participate in the study and sign an Informed Consent Form;
2. Female subjects aged 18 years or older at the time of signing the Informed Consent Form;
3. Histology confirmed high grade serous ovarian, fallopian tube or primary peritoneal cancer;
4. Must be newly developed platinum-resistant (Must not have received systemic therapy after developing platinum resistance status);
5. Received at least 3 prior lines of systemic therapies；
6. Imaging evidence of disease progression during or at the end of last-line therapy;
7. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1;
8. Life expectancy of at least 12 weeks;
9. Subjects are willing to provide archival tumor tissue samples or accept a low-risk routine medical procedure to collect the fresh biopsy sample for immunohistochemical (IHC) MSLN testing;
10. Measurable lesion according to RECIST v1.1；
11. The interval between previous focal radiotherapy and the first dose should be at least 2 weeks；
12. Have laboratory tests that meet the relevant requirements to demonstrate adequate organ function;
13. Subjects of childbearing potential are required to use effective contraception from the time of informed consent and continuing through 6 months after the final dose of study intervention; Fertile subjects included those who were not menopausal or had been menopausal for less than 2 years and had not undergone bilateral adnexectomy or hysterectomy；Subjects of childbearing potential must have a negative pregnancy test within 7 days prior to the first dose of study intervention.

Exclusion Criteria:

1. The presence of clinically uncontrollable third-space fluids, such as massive pleural effusion or pericardial effusion accompanied by clinical symptoms or requiring symptomatic management; and ascites that cannot be effectively controlled with treatment;
2. Subjects with asymptomatic brain metastases who have received prior treatment may participate in this study if they meet all the following criteria:

   * Only supratentorial and/or cerebellar metastases are present.
   * Corticosteroids should be discontinued for at least 7 days prior to the first dose;
   * No disease progression is observed on imaging from completion of brain-directed therapy until randomization compared to pre-treatment imaging (at least 4 weeks interval).
   * Subjects must undergo radiotherapy and/or surgery for brain metastases if new asymptomatic brain metastases are detected during screening period.
3. Subjects with a history of other invasive malignancies within 3 years prior to the first dose, except for adequately treated papillary thyroid carcinoma, basal cell or squamous cell skin cancers without evidence of recurrence, and other adequately treated carcinoma in situ without evidence of disease recurrence；
4. Subjects with ongoing clinically significant toxicity associated with prior treatment that has not resolved to Grade 0 or 1 by NCI CTCAE 5.0;
5. Subjects who have received systemic anti-tumor therapy (including chemotherapy, targeted therapy, biologic therapy, hormonal therapy, etc.) within 28 days or 5 half-lives of prior therapy (whichever is shorter) prior to first dose;
6. Subjects who have received herbal or proprietary Chinese medicines for tumor control within 14 days prior to the first dose;
7. Subjects who have received previous mesothelin target-related drugs or MMAE, MMAF, DM1, DM4 and other microtubule inhibitor ADCs；
8. Subjects with clinical symptoms or signs of gastrointestinal obstruction;
9. History of cirrhotic liver disease (Child-Pugh Class B or C);
10. Subjects with immunodeficiency diseases, currently receiving systemic glucocorticoid therapy (dose>10 mg/d of prednisone or equivalent dose among drugs in the same class), or receiving immune suppressant therapy within 7 days prior to the first dose；
11. Major surgery within 4 weeks and no fully recovered prior to the first dose or anticipation of surgery；
12. Patients with active or progressive infection that requiring systemic therapy within 14 days prior to first dose, such as active tuberculosis;
13. serum virological testing (based on study center normal values)

    * Positive results of Hepatitis B virus surface antigen (HBsAg) should be further tested for HBV DNA, HBV DNA > 200IU/ml or 2000 copies /ml cannot be enrolled. However, if subjects received nucleotide-based antiviral therapy and test result below the criteria above, they could be enrolled;
    * Positive results of Hepatitis C antibody (HCVAb) (HCV RNA>103 copies/ml) cannot be enrolled. However, if subjects received nucleotide-based antiviral therapy and the test result below the criteria above, they could be enrolled;
    * Positive results for human immunodeficiency virus antibody (HIVAb).
14. Subjects with prior allogeneic haematopoietic stem cell transplantation or solid organ transplantation, or those who are waiting for organ transplantation;
15. Uncontrolled or significant cardiovascular and cerebrovascular diseases;
16. A history of interstitial lung disease requiring treatment or currently having a severe pulmonary disease, including but not limited to interstitial lung disease;
17. In the investigator's opinion, any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory findings, that raise reasonable suspicion of a disease or condition affecting the interpretation of the study results or placing the patient at high risk of participating in the study；
18. Subjects with active corneal disease and those who, in the judgement of the ophthalmologist, are unsuitable for inclusion by funduscopic examination and other ocular related examinations；
19. Subjects with known allergies to RC88 or its excipients or have had a history of severe allergic reactions to the other monoclonal antibodies or chemotherapies;
20. Subjects who have received a live or live-attenuated vaccine within 4 weeks prior to the first dose or plan to receive the above vaccines during the study；
21. Known psychiatric or substance abuse disorders that may have an impact on compliance with the study requirements.
22. Pregnant and/or breast-feeding women；
23. The subject's compliance are estimated to be insufficient to participate in this study, or other factors that, in the investigator's opinion, make the subjects unsuitable for participation of this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2024-01-19 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) by Independent Review Committee (IRC) | Up to approximately 2 years
  The proportion of subjects whose BOR is a confirmed CR or PR. Tumor response will be evaluated by IRC using RECIST v.1.1.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) by investigator | Up to approximately 2 years
  The proportion of subjects whose BOR is a confirmed CR or PR. Tumor response will be evaluated by investigator using RECIST v.1.1.
Duration of response (DOR) by Independent Review Committee (IRC) | Up to approximately 2 years
  The duration from first documentation of response (CR or PR) until the time of first documentation of disease progression or death. Tumor response will be evaluated by IRC using RECIST v.1.1.
Duration of response (DOR) by investigator | Up to approximately 2 years
  The duration from first documentation of response (CR or PR) until the time of first documentation of disease progression or death. Tumor response will be evaluated by the investigator using RECIST v.1.1.
Progression-free survival (PFS) by Independent Review Committee (IRC) | Up to approximately 2 years
  The duration from first dose to disease progression or death as assessed by IRC using RECIST v1.1 criteria.
Progression-free survival (PFS) by investigator | Up to approximately 2 years
  The duration from first dose to disease progression or death as assessed by the investigator using RECIST v1.1 criteria.
Overall survival (OS) | Up to approximately 2 years
  The duration from the date of the first dose of study treatment to the date of death.
CA-125 relieve defined by GCIG | Up to approximately 2 years
  Serum CA125 Assessment defined by GCIG
The peak and trough concentrations of RC88 binding antibody (ADC), total antibody (TAb) and free MMAE | Up to approximately 2 years
  The peak and trough concentrations of RC88 binding antibody (ADC), total antibody (TAb) and free MMAE will be detected.
Incidence of Anti-Drug Antibodies (ADA), titers, and/or neutralizing antibodies (NAb) Rate etc. | Up to approximately 2 years
  Incidence of Anti-Drug Antibodies (ADA), titers, and/or neutralizing antibodies (NAb) Rate etc.will be detected.
Safety: The types, incidence, correlation, and severity of various adverse events (AES), as well as the types, incidence, and severity of laboratory abnormalities | Up to approximately 2 years
  The types, incidence, correlation, and severity of various adverse events (AES), as well as the types, incidence, and severity of laboratory abnormalities will be detected.

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, M.D, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Beihua Kong, M.D, Principal Investigator — Qilu Hospital of Shandong University; Jie Jiang, M.D, Principal Investigator — Qilu Hospital of Shandong University
Locations (30):
- China (30):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Xingtai People's Hospital, Xingtai, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shandong Cancer Hospital, Shandong Cancer Institute, Jinan, Shandong
  - Qingdao Central Hospital, Qingdao, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shangdong
  - Obstetrics & Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Second hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The West China Second University Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No